CLINICAL TRIAL: NCT00979420
Title: Non-interventional Observational Study With Viramune (Nevirapine) and Various Drug Combinations in the Antiretroviral Combination Treatment of HIV-infected Patients Who Have Already Been Treated for Approx. 10 Years With Viramune
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1100.1535
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: HIV Infections
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HIV treatment

SUMMARY:
The question that prompted this study is the extent to which results from clinical trials can be translated into everyday practice (external validity). An observation period of about 10 years extends far beyond the duration of clinical trials. First and foremost are questions about tolerability and the efficacy of an antiretroviral combination treatment with Viramune and other antiretroviral partners. In particular, adverse events will be recorded and the therapeutic effect will be monitored via the course of viral load and improvement of the immune system, based on the CD4 cell count.

DETAILED DESCRIPTION:
Study Design:

observational

ELIGIBILITY:
Inclusion criteria The inclusion criteria for treatment with Viramune plus other antiretroviral combination drugs are to be based on the current Information for Healthcare Professionals/SPC (R08-0843)

Exclusion criteria The exclusion criteria for treatment with Viramune plus other antiretroviral combination drugs are to be based on the current Information for Healthcare Professionals/SPC (R08-0843).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Dates: Start 2009-08; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (60):
- Germany (60):
  - Boehringer Ingelheim Investigational Site 1, Aachen
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 15, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 16, Bochum
  - Boehringer Ingelheim Investigational Site 17, Bonn
  - Boehringer Ingelheim Investigational Site 18, Bremen
  - Boehringer Ingelheim Investigational Site 19, Dortmund
  - Boehringer Ingelheim Investigational Site 20, Duisburg
  - Boehringer Ingelheim Investigational Site 21, Düsseldorf
  - Boehringer Ingelheim Investigational Site 22, Düsseldorf
  - Boehringer Ingelheim Investigational Site 23, Düsseldorf
  - Boehringer Ingelheim Investigational Site 24, Düsseldorf
  - Boehringer Ingelheim Investigational Site 25, Frankfurt
  - Boehringer Ingelheim Investigational Site 26, Frankfurt
  - Boehringer Ingelheim Investigational Site 27, Frankfurt
  - Boehringer Ingelheim Investigational Site 28, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 29, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 30, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 31, Hamburg
  - Boehringer Ingelheim Investigational Site 32, Hamburg
  - Boehringer Ingelheim Investigational Site 33, Hamburg
  - Boehringer Ingelheim Investigational Site 34, Hamburg
  - Boehringer Ingelheim Investigational Site 35, Hamburg
  - Boehringer Ingelheim Investigational Site 36, Hamburg
  - Boehringer Ingelheim Investigational Site 37, Hanover
  - Boehringer Ingelheim Investigational Site 38, Hanover
  - Boehringer Ingelheim Investigational Site 39, Hanover
  - Boehringer Ingelheim Investigational Site 40, Heidelberg
  - Boehringer Ingelheim Investigational Site 41, Karlsruhe
  - Boehringer Ingelheim Investigational Site 42, Koblenz
  - Boehringer Ingelheim Investigational Site 43, Leipzig
  - Boehringer Ingelheim Investigational Site 44, Mannheim
  - Boehringer Ingelheim Investigational Site 45, Mannheim
  - Boehringer Ingelheim Investigational Site 46, München
  - Boehringer Ingelheim Investigational Site 47, München
  - Boehringer Ingelheim Investigational Site 48, München
  - Boehringer Ingelheim Investigational Site 49, München
  - Boehringer Ingelheim Investigational Site 50, München
  - Boehringer Ingelheim Investigational Site 51, Münster
  - Boehringer Ingelheim Investigational Site 52, Münster
  - Boehringer Ingelheim Investigational Site 53, Münster
  - Boehringer Ingelheim Investigational Site 54, Oldenburg
  - Boehringer Ingelheim Investigational Site 55, Osnabrück
  - Boehringer Ingelheim Investigational Site 56, Saarbrücken
  - Boehringer Ingelheim Investigational Site 57, Stuttgart
  - Boehringer Ingelheim Investigational Site 58, Stuttgart
  - Boehringer Ingelheim Investigational Site 59, Stuttgart
  - Boehringer Ingelheim Investigational Site 60, Wuppertal

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment-naive Patients: Patient was not treated with any antiretroviral drugs (ARV) before start of therapy with Viramune
- Pre-treated Patients With Baseline HIV RNA <50 Copies/ml: HIV RNA denotes Human immunodeficiency virus (HIV) Ribonucleic acid (RNA). Baseline reflects the last available documentation before start of treatment with Viramune
- Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml; Pre-treated Patients With Baseline HIV RNA Not Documented: Baseline reflects the last available documentation before start of treatment with Viramune
Period: Overall Study
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA <50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Started | 178 | 57 | 60 | 61
Completed | 171 | 57 | 59 | 59
Not Completed | 7 | 0 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 1 | 1
Not completed — Other reasons not related to Viramune | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set - all patients receiving at least one dose of study medication
Groups:
- Pre-treated Patients With Baseline HIV RNA<50 Copies/ml; Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml; Pre-treated Patients With Baseline HIV RNA Not Documented: Baseline reflects the last available documentation before start of treatment with Viramune
- Total: Total of all reporting groups
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented | Total
Number analyzed (Participants) | 178 | 57 | 60 | 61 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.85 (10.54) | 54.21 (10.42) | 51.02 (7.66) | 53.69 (11.05) | 51.91 (10.24)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 142 | 44 | 41 | 51 | 278
  Female | 36 | 13 | 19 | 9 | 77
  Missing | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in log10 Viral Load From Baseline to Last Visit
Description: Baseline is defined as the last documentation before start of therapy with Viramune. The change from baseline reflects the last available visit viral load minus the baseline viral load.
Time Frame: Baseline and last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: Full analysis set (FAS): This patient set includes all patients from Treated Set (TS) who have documented at least one value for the viral load before start of therapy with Viramune.
Measure: Median (Full Range); unit: log10 copies/ml
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 86 | 57 | 60
log10 copies/ml | -3.260 (-5.61;2.25) [-5.61 to 2.25] | -0.099 (-1.69;0.70) [-1.69 to 0.70] | -2.082 (-5.82;0.40) [-5.82 to 0.40]

2. Primary Outcome: Number of Participants With Viral Load <50 Copies/ml and >=50 Copies/ml at Last Visit
Time Frame: Last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: FAS: This patient set includes all patients from TS who have documented at least one value for the viral load before start of therapy with Viramune.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 86 | 57 | 60
Participants
  <50 copies/ml | 83 | 55 | 55
  >=50 copies/ml | 3 | 2 | 5
  Missing | 0 | 0 | 0

3. Primary Outcome: Change in Absolute CD4 Lymphocytes (CD4+) Cells From Baseline to Last Visit
Description: Baseline is defined as the last documentation before start of therapy with Viramune. The change from baseline reflects the last available number of CD4+ cells minus the baseline number of CD4+ cells.
Time Frame: Baseline and last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: as for outcome 2
Measure: Median (Full Range); unit: CD4+ cells/mm3
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 83 | 56 | 60
CD4+ cells/mm3 | 380 (-323;1749) [-323 to 1749] | 223.5 (-328;1104) [-328 to 1104] | 228 (-360;1004) [-360 to 1004]

4. Primary Outcome: Change in log10 Viral Load From Baseline to Last Visit
Description: as for outcome 1
Time Frame: Baseline and last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: Per protocol set (PPS): All patients from FAS without treatment interruptions and who are treated with Viramune for at least 10 years.
Measure: Median (Full Range); unit: log10 copies/ml
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 63 | 34 | 33
log10 copies/ml | -3.284 (-5.61;0.00) [-5.61 to 0.00] | 0.000 (-0.41;0.70) [-0.41 to 0.70] | -2.000 (-5.824;0.40) [-5.824 to 0.40]

5. Primary Outcome: Number of Participants With Viral Load <50 Copies/ml and >=50 Copies/ml at Last Visit
Time Frame: Last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: PPS: All patients from FAS without treatment interruptions and who are treated with Viramune for at least 10 years.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 63 | 34 | 33
Participants
  <50 copies/ml | 62 | 33 | 30
  >=50 copies/ml | 1 | 1 | 3

6. Primary Outcome: Change in Absolute CD4 Lymphocytes (CD4+ Cells) From Baseline to Last Visit
Description: as for outcome 3
Time Frame: Baseline and last available visit. Duration of intake of Viramune ranges from 14 to 185 months.
Population: PPS: All patients from FAS without treatment interruptions and who are treated with Viramune for at least 10 years.
Measure: Median (Full Range); unit: CD4+ cells/mm3
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 61 | 33 | 33
CD4+ cells/mm3 | 392 (-323;1027) [-323 to 1027] | 283 (-234;1104) [-234 to 1104] | 250 (-266;987) [-266 to 987]

7. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Cholesterol During Study (Worst Grade) by Division of AIDS (DAIDS) Grade
Description: Duration of intake of Viramune ranges from 14 to 185 months. The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("DAIDS AE Grading Table") was used for grading the safety laboratory parameters. Grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = potentially life-threatening.
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of cholesterol.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 90 | 28 | 21 | 37
Participants
  < Grade 1 | 11 | 7 | 4 | 2
  Grade 1 | 26 | 8 | 4 | 18
  Grade 2 | 40 | 10 | 9 | 8
  Grade 3 | 13 | 3 | 4 | 9
  Grade 4 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Low-density Lipoprotein (LDL) Cholesterol During Study (Worst Grade) by DAIDS Grade
Description: Duration of intake of Viramune ranges from 14 to 185 months. The "DAIDS AE Grading Table" was used for grading the safety laboratory parameters. Grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = potentially life-threatening.
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of LDL cholesterol.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 76 | 23 | 18 | 33
Participants
  < Grade 1 | 17 | 9 | 5 | 9
  Grade 1 | 30 | 6 | 5 | 8
  Grade 2 | 11 | 5 | 3 | 13
  Grade 3 | 18 | 3 | 5 | 3
  Grade 4 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Triglycerides During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of triglycerides.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 91 | 28 | 21 | 37
Participants
  < Grade 1 | 72 | 27 | 17 | 26
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 15 | 1 | 2 | 4
  Grade 3 | 3 | 0 | 1 | 4
  Grade 4 | 1 | 0 | 1 | 3

10. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Blood Glucose During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of blood glucose
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 175 | 57 | 59 | 59
Participants
  < Grade 1 | 50 | 22 | 21 | 12
  Grade 1 | 83 | 25 | 25 | 25
  Grade 2 | 29 | 5 | 7 | 17
  Grade 3 | 8 | 1 | 1 | 3
  Grade 4 | 5 | 4 | 5 | 2

11. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Alanine Aminotransferase (ALT) During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of ALT
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 59 | 58
Participants
  < Grade 1 | 94 | 32 | 27 | 28
  Grade 1 | 68 | 17 | 27 | 22
  Grade 2 | 12 | 7 | 3 | 4
  Grade 3 | 4 | 1 | 1 | 2
  Grade 4 | 0 | 0 | 1 | 2

12. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Aspartate Aminotransferase (AST) During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of AST
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 59 | 58
Participants
  < Grade 1 | 105 | 40 | 40 | 30
  Grade 1 | 58 | 12 | 14 | 20
  Grade 2 | 12 | 5 | 3 | 7
  Grade 3 | 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 1 | 1

13. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Creatinine During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of Creatinine.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 60 | 59
Participants
  < Grade 1 | 152 | 51 | 50 | 49
  Grade 1 | 13 | 3 | 5 | 3
  Grade 2 | 2 | 0 | 2 | 1
  Grade 3 | 1 | 0 | 0 | 1
  Grade 4 | 10 | 3 | 3 | 5

14. Secondary Outcome: Number of Patients With Laboratory Abnormalities for Hemoglobin During Study (Worst Grade) by DAIDS Grade
Description: as for outcome 8
Time Frame: Up to 185 months
Population: Patients from Treated set (TS, all patients receiving at least one dose of study medication) with at least one documentation of Hemoglobin.
Measure: Number; unit: Participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA<50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 56 | 60 | 59
Participants
  < Grade 1 | 171 | 53 | 58 | 54
  Grade 1 | 6 | 1 | 1 | 3
  Grade 2 | 1 | 2 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 1 | 2

15. Secondary Outcome: Duration of Intake of Viramune
Description: Duration of intake of Viramune
Time Frame: End of treatment, up to 185 months
Population: Treated set
Measure: Median (Full Range); unit: months
Groups:
- Pre-treated Patients With Baseline HIV RNA <50 Copies/ml; Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml; Pre-treated Patients With Baseline HIV RNA Not Documented: Baseline reflects the last available documentation before start of treatment with Viramune
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA <50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 60 | 61
months | 131 [30 to 185] | 124 [43 to 149] | 131 [14 to 159] | 129 [105 to 161]

16. Secondary Outcome: History of Therapy With Antiretroviral Medication
Description: Participants with a history of therapy with antiretroviral medication.
Time Frame: Baseline
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA <50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 60 | 61
participants
  Treatment-naive | 178 | 0 | 0 | 0
  Pre-treated | 0 | 57 | 60 | 61

17. Secondary Outcome: Course of Absolute CD4+ Cell Count
Description: The course of absolute CD4+ cell count is presented as the absolute CD4+ cell count at last visit.
Time Frame: Baseline and last available visit. Duration of intake of Viramune ranges from 14 to 185 months
Population: PPS: All patients from FAS without treatment interruptions and who are treated with Viramune for at least 10 years
Measure: Median (Full Range); unit: CD4+ cells/mm3
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA <50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml
Number analyzed (Participants) | 63 | 33 | 33
CD4+ cells/mm3 | 734 [96 to 1526] | 669 [189 to 1479] | 491 [237 to 1326]

18. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: Number of participants with drug related Adverse Events (AEs)
Time Frame: Up to 185 months
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Pre-treated Patients With Baseline HIV RNA <50 Copies/ml | Pre-treated Patients With Baseline HIV RNA>=50 Copies/ml | Pre-treated Patients With Baseline HIV RNA Not Documented
Number analyzed (Participants) | 178 | 57 | 60 | 61
participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 14 to 185 months
Arm/Group | Viramune
Serious Adverse Events (participants affected / at risk) | 35/356
Other Adverse Events (participants affected / at risk) | 60/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viramune (N=356)
Acute myocardial infarction (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac valve disease (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery occlusion (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 8
Abdominal pain lower (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 2
Pneumonia pneumococcal (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1
Substance abuse (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Caesarean section (Surgical and medical procedures) | 7
Venous thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Viramune (N=356)
Diarrhoea (Gastrointestinal disorders) | 21
Bronchitis (Infections and infestations) | 20
Hypertension (Vascular disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.